CLINICAL TRIAL: NCT01046396
Title: Split-Face Tolerability Comparison Between Differin® Cream 0.1% Versus Differin® Lotion 0.1% in Subjects With Healthy Skin
Brief Title: Tolerability Comparison of Differin® Cream 0.1% Versus Differin® Lotion 0.1% in Subjects With Healthy Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10149
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2012-09

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Differin® Cream 0.1% (Active Comparator): Adapalene Cream 0.1% - apply once daily on one side of the face for 3 weeks
  Interventions: Drug: adapalene cream 0.1% and adapalene lotion 0.1%
- Differin® Lotion 0.1% (Active Comparator): Adapalene Lotion 0.1% - apply once daily on the opposite side of the face for 3 weeks
  Interventions: Drug: adapalene lotion 0.1%

INTERVENTIONS:
Drug: adapalene cream 0.1% and adapalene lotion 0.1% — adapalene cream 0.1% - apply once daily on one side of the face for 3 weeks
  Other Names: Differin® Cream 0.1%
  Arms: Differin® Cream 0.1%
Drug: adapalene lotion 0.1% — adapalene lotion 0.1% - apply once daily on the opposite side of the face for 3 weeks
  Other Names: Differin® Lotion 0.1%
  Arms: Differin® Lotion 0.1%

SUMMARY:
The purpose of this study is to compare the tolerability of Differin® (adapalene) Cream, 0.1% to Differin® Lotion, 0.1% in subjects with healthy skin treated once a day for three (3) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years and older
* Subjects with healthy skin as determined by the clinical grader

Exclusion Criteria:

* Subjects with a degree of skin pigmentation that interferes with the reading of skin reactions.
* Subjects with a condition or who are in a situation, which in the investigator's opinion may put the subject at risk, may confound study results, or may interfere with the subject's participation in the study.
* Subjects with known allergy to one of the components of the study drugs (refer to the package insert for Differin® Cream 0.1% and the investigator's brochure for Differin® Lotion 0.1%).
* Subjects who have participated in another investigational drug or device research study within 30 days of enrollment.
* Subjects with a washout period for topical treatment on the treated area less than 1 week for corticosteroids and/or 4 weeks for retinoids.
* Subjects with a washout period for systemic treatment less than 1 week for medications that may increase photosensitivity and/or 4 weeks for corticosteroids and/or 6 months for retinoids.
* Subjects with current sunburn, eczema, atopic dermatitis, perioral dermatitis or rosacea on the area to be treated.
* Subjects who foresee unprotected and intense UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Thomas J. Stephens & Associates, Inc., Colorado Springs, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: First subject was enrolled on January 11, 2010 and the last subject was enrolled on January 13, 2010.
  Types of location: Investigative site was located at a research center.
Pre-assignment Details: Wash-out period up to baseline for topical treatment on the treated area was less than 1 week for corticosteroids and/or 4 weeks for retinoids; for systemic treatment, it was less than 1 week for medications that may have increased photosensitivity and/or 4 weeks for corticosteroids and/or 6 months for retinoids.
Groups:
- Differin® Cream 0.1% and Differin® Lotion 0.1%: Adapalene Cream 0.1% - apply topically to one side of the face once daily for 3 weeks; Adapalene Lotion 0.1% - apply to the opposite side of the face for 3 weeks
Period: Overall Study
Arm/Group | Differin® Cream 0.1% and Differin® Lotion 0.1%
Started | 69
Completed | 64
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Differin® Cream 0.1% and Differin® Lotion 0.1%
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.87 (13.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were a Success With Regard to Worst Post-baseline Tolerability Assessment Scores in Each Category of the Tolerability Assessments (Erythema, Scaling, Dryness, Stinging/Burning) From Baseline to Week 3.
Description: Number of participants who were a success with regard to worst post-baseline tolerability assessment scores in each category of the tolerability assessments from baseline to week 3. Tolerability assessments (erythema, scaling, dryness, stinging/burning) are evaluated on a scale from 0 - 4 (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe) with 0 being best and 4 being worst. Success for each category was defined as a tolerability score of 0.
Time Frame: baseline to week 3
Population: Per protocol
Measure: Number; unit: participants
Groups:
- Differin® Cream 0.1%: Adapalene Cream 0.1% - apply topically to one side of the face once daily for 3 weeks
- Differin® Lotion 0.1%: Adapalene Lotion 0.1% - apply to the opposite side of the face for 3 weeks
Arm/Group | Differin® Cream 0.1% | Differin® Lotion 0.1%
Number analyzed (Participants) | 64 | 64
participants
  Erythema | 9 | 9
  Scaling | 32 | 30
  Dryness | 14 | 14
  Stinging / Burning | 58 | 56

2. Secondary Outcome: 6 Question Subject Cosmetic Acceptability Questionnaire at Week 3
Description: Number of participants in each category (Differin® Lotion, Differin® Cream or No Preference) of each question of the Subject Cosmetic Acceptability Questionnaire at week 3.
Time Frame: week 3
Population: ITT (Intent to Treat)
Measure: Number; unit: participants
Groups:
- No Preference: Neither Differin® Cream 0.1% nor Differin® Lotion 0.1%
Arm/Group | Differin® Cream 0.1% | Differin® Lotion 0.1% | No Preference
Number analyzed (Participants) | 69 | 69 | 69
participants
  Which side was easier to apply? | 19 | 12 | 33
  Which side absorbed into your skin more quickly? | 27 | 17 | 20
  Which side had less odor? | 7 | 10 | 47
  Which side felt better on your skin? | 26 | 15 | 23
  Which side left less residue on your skin? | 18 | 15 | 31
  Generally, which side did you prefer? | 23 | 13 | 28

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Subjects were asked if there had been any change in their health at each study visit; information obtained was recorded as adverse event(s), when applicable.
Arm/Group | Differin® Cream 0.1% | Differin® Lotion 0.1%
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 5/69 | 5/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Differin® Cream 0.1% (N=69) | Differin® Lotion 0.1% (N=69)
head cold (Infections and infestations) | 5 (5) | 5 (5) — The subjects in the Differin® Cream arm who experienced a head cold were the same as the subjects who experienced a head cold in the Differin® Lotion arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator has the right to publish or present the data resulting from this study, with agreed upon reviews by all interested parties, and in accordance with any confidentiality agreements that may exist.